CLINICAL TRIAL: NCT00136045
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Four-arm Parallel-group Trial to Investigate the Efficacy and Safety of Three Different Transdermal Doses of Rotigotine in Subjects With Idiopathic Restless Leg Syndrome
Brief Title: Three Different Transdermal Doses of Rotigotine in Subjects With Idiopathic Restless Leg Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0790; 2005-000428-18 (EudraCT Number)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2010-02

CONDITIONS: Restless Legs Syndrome
Keywords: Idiopathic RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
The primary objective of this trial is to demonstrate that rotigotine (SPM 936) is efficacious in subjects with idiopathic restless leg syndrome (RLS). Additional objectives are to investigate the safety and tolerability of rotigotine.

The primary variables are the absolute change from Baseline in the International Restless Legs Severity Scale (IRLS) sum score and Clinical Global Impression-Global Improvement (CGI) Item 1 (severity of illness) score at the end of the Maintenance Period.

Subjects will be randomized to receive either placebo, 2.25, 4.5 or 6.75 mg/day rotigotine in a 1:1:1:1 (active:placebo) fashion. Approximately 450 subjects will be enrolled in this trial, participating at approximately 50 sites. The maximum duration of the trial is approximately 8 months (3-week Titration Period, 6-month Maintenance Period, 7-day Taper Period, and 30-day Safety Follow-Up Period). Subjects who complete the 6-month Maintenance Period will be eligible to participate in an open-label extension trial. Subjects who do not complete the 6-month Maintenance Period or who choose not to participate in the open-label extension trial will complete a 3-day Safety Follow-Up Period. Two different patch sizes will be used (5 and 10 cm2). Active patches will contain either 2.25mg (5cm2) or 4.5mg (10cm2) of rotigotine.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic RLS

Exclusion Criteria:

* History of sleep disturbances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2005-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
IRLS sum score and CGI Item 1 score severity of illness | From Baseline at the end of the Maintenance Period

SECONDARY OUTCOMES:
IRLS Responder: A responder is a subject with a decrease of ≥50% in IRLS sum score from Baseline at the end of the Maintenance Period
Changes in CGI Items 2-3 (continuous) during the Maintenance Period; Change from Baseline in RLS-6 Rating Scales at the end of the Maintenance Period
CGI Item 1 Responder: A responder is a subject with a decrease of ≥50% in CGI Item 1 at the end of the Maintenance Period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Trenkwalder C, Benes H, Poewe W, Oertel WH, Garcia-Borreguero D, de Weerd AW, Ferini-Strambi L, Montagna P, Odin P, Stiasny-Kolster K, Hogl B, Chaudhuri KR, Partinen M, Schollmayer E, Kohnen R; SP790 Study Group. Efficacy of rotigotine for treatment of moderate-to-severe restless legs syndrome: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2008 Jul;7(7):595-604. doi: 10.1016/S1474-4422(08)70112-1. PMID 18515185
- [Derived] Ondo WG, Grieger F, Moran K, Kohnen R, Roth T. Post Hoc Analysis of Data from Two Clinical Trials Evaluating the Minimal Clinically Important Change in International Restless Legs Syndrome Sum Score in Patients with Restless Legs Syndrome (Willis-Ekbom Disease). J Clin Sleep Med. 2016 Jan;12(1):63-70. doi: 10.5664/jcsm.5396. PMID 26446245
- [Derived] Allen R, Oertel W, Walters A, Benes H, Schollmayer E, Grieger F, Moran K, Kohnen R. Relation of the International Restless Legs Syndrome Study Group rating scale with the Clinical Global Impression severity scale, the restless legs syndrome 6-item questionnaire, and the restless legs syndrome-quality of life questionnaire. Sleep Med. 2013 Dec;14(12):1375-80. doi: 10.1016/j.sleep.2013.09.008. Epub 2013 Oct 18. PMID 24246378